CLINICAL TRIAL: NCT00221975
Title: Combination Therapy in Dual Diagnosis Rapid Cycling Bipolar Disorder
Brief Title: Combination Therapy in Dual Diagnosis Bipolar Rapid Cycling
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Joseph Calabrese, MD, Director, Mood Disorders Program, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 02T 183
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Valproic Acid; Lamotrigine; Lithium; Lithium Carbonate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lithium + Divalproex + Lamictal (Active Comparator): Lithium monotherapy was initiated at 450 mg once daily and titrated slowly over 3 weeks to a minimum blood level of 0.5 mEqlL. Divalproex was then initiated at 250 mg twice daily and increased slowly over 5 weeks to a minimum blood level of 50 μg/mL. Patients meeting the criteria of being non-responsive to lithium plus divalproex were randomly assigned to receive lamotrigine or placebo. Patients randomized to the lamotrigine group were titrated up to a minimum dose of 150 mg and maximum dose of 200 mg per day.
  Interventions: Drug: Divalproex; Drug: Lamotrigine; Drug: Lithium
- Lithium + Divalproex + Placebo (Placebo Comparator): Lithium monotherapy was initiated at 450 mg once daily and titrated slowly over 3 weeks to a minimum blood level of 0.5 mEqlL. Divalproex was then initiated at 250 mg twice daily and increased slowly over 5 weeks to a minimum blood level of 50 μg/mL. Patients meeting the criteria of being non-responsive to lithium plus divalproex were randomly assigned to receive lamotrigine or placebo. Patients randomized to the placebo group were giving matching placebo.
  Interventions: Drug: Divalproex; Drug: Lithium

INTERVENTIONS:
Drug: Divalproex — Once a therapeutic blood level of lithium was achieved, Divalproex was initiated at 250 mg twice daily and increased slowly over 5 weeks to a minimum blood level of 50 μg/mL.
  Other Names: Depakote
Drug: Lamotrigine — Lithium monotherapy was initiated at 450 mg once daily and titrated slowly over 3 weeks to a minimum blood level of 0.5 mEqlL.
  Other Names: Lamictal
  Arms: Lithium + Divalproex + Lamictal
Drug: Lithium — Subjects who did not respond to the combination of Lithium and Divalproex were then randomly assigned in a 1:1 ratio to adjunctive lamotrigine versus placebo after stratification by illness type (bipolar I versus bipolar II), historical response to lithium (response versus oon-response), and the length of current exposure to the combination treatment with lithium and divalproex (<2 months versus ≥2 months).
  Other Names: Eskalith

SUMMARY:
Combination Therapy in Dual Diagnosis Bipolar Rapid Cycling: This study recruits males and females age 18 and older who currently meet diagnostic criteria for rapid cycling bipolar disorder (type I or II) and who have met the criteria for substance abuse or dependence of cocaine, marijuana and/or alcohol within the past six months. Patients begin treatment with a combination of lithium and divalproex. Once these medications are tolerated, they are randomly assigned to double-blind treatment with lamotrigine or placebo. Patients remain in this study until they experience a marked bimodal response for four consecutive weeks. This study is sponsored by the Stanley Foundation.

ELIGIBILITY:
Inclusion Criteria:

* Has given written informed consent.
* Males or females 16 years of age and older. For patients less than 18 years old, concurrent written informed consent will also be required from the parents or legal guardians.
* Must meet Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria for major depression at the time of study entry.
* Must meet DSM-IV criteria for rapid-cycling bipolar disorder in the last 12 months.
* Must meet DSM-IV criteria for alcohol or drug abuse within the past 3 months or dependence in the last 6 months (unless most recent period of abstinence occurred while in a controlled environment).
* Must have no medical illness precluding the use of lithium, divalproex sodium and/or lamotrigine.
* Regardless of treatment response, patients who have been exposed to lithium or divalproex sodium will be included as long as the medication was adequately tolerated and all three medications were not administered concurrently.

Exclusion Criteria:

* Patients who have had intolerable side effects to lamotrigine, lithium at levels of 0.6 mEq/L or divalproex sodium at levels of 50ug/ml.
* Patients who have previously been treated with lithium, divalproex sodium and lamotrigine concurrently.
* Patients who have previously been treated with an adequate trial of lamotrigine, which was considered to be a treatment failure.
* Patients who do not have a recent history of, or are not currently abusing or dependent on alcohol or drugs.
* Patients with a prior history of seizure disorder, cerebral vascular disease, structural brain damage from trauma, clinically significant focal neurological abnormalities, closed head injury, EEG abnormalities with frank paroxysmal activity or a previous CT/MRI scan of the brain with gross structural abnormalities.
* Patients who have clinically significant gastrointestinal, renal, hepatic, endocrine, cardiovascular, pulmonary, immunologic, hematologic, or oncologic diseases. Clinically significant evidence of thyroid failure will be defined as a decreased free thyroxine index with several clinical signs and symptoms of overt failure.
* Patients who are pregnant, at-risk of becoming pregnant or intend to become pregnant during the study. Patients who are not at risk of becoming pregnant are females who are post menopausal, who have undergone a hysterectomy, bilateral oophorectomy or sterilization, who agree to use an IUD, barrier protection, a contraceptive implantation system (e.g., Norplant), oral contraceptive pills, or who, in the investigator's judgment, will continue to be sexually inactive.
* Patients who have received haloperidol decanoate or fluphenazine decanoate within the last 10 weeks.
* Patients who have a central nervous system (CNS) neoplasm, uncontrolled metabolic, demyelinating or progressive degenerative disorder, active CNS infection, or any progressive neurological disorder.
* Patients who are taking exogenous steroids.
* Patients who have ultra-fast rapid-cycling bipolar disorder, but do not formally meet DSM-IV criteria for bipolar disorder. This is designed to exclude patients with episode frequencies too high to permit objective quantification.
* Patients who are currently suicidal in the opinion of the investigator or have a score of greater than 4 on the suicide item of the (Montgomery-Asberg Rating Scale (MADRS).
* Patients who have been treated with any dose or duration of a tricyclic antidepressant within the last three months.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2002-07; Primary Completion 2007-06 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who experience a marked and persistent bimodal response | Phase 1: Baseline - Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Keming Gao, MD, PhD, Principal Investigator — Case Western Reserve University / University Hospitals of Cleveland
Locations (1):
- University Hospitals of Cleveland, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Gao K, Verduin ML, Kemp DE, Tolliver BK, Ganocy SJ, Elhaj O, Bilali S, Brady KT, Findling RL, Calabrese JR. Clinical correlates of patients with rapid-cycling bipolar disorder and a recent history of substance use disorder: a subtype comparison from baseline data of 2 randomized, placebo-controlled trials. J Clin Psychiatry. 2008 Jul;69(7):1057-63. doi: 10.4088/jcp.v69n0703. PMID 18588360